CLINICAL TRIAL: NCT00569907
Title: Observational Study of Interstitial Glucose Monitoring With Continuous Glucose Monitoring to Track Patients Treated With Exenatide
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Roger S. Mazze, PhD - Chief Academic Officer, Park Nicollet Institute dba International Diabetes Center
Other Study IDs: 03520-06-C
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus Type 2
Keywords: type 2 diabetes; continuous glucose monitoring; exenatide; exenatide use
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Approximately 30 adults will participate in this study at the International Diabetes Center (IDC). The IDC is the only site conducting this study.

Length of participation can range from two to three months which will include four to seven clinic visits.

The purpose of this study is to use a Continuous Glucose Monitoring (CGM) system to determine the characteristics of glucose control and patterns of food intake before exenatide is started, during the start and adjustment of exenatide and during exenatide treatment.

The long-term purpose of this study is to determine to what extent continuous glucose monitoring improves or alters clinical decision making for patients treated with exenatide. And, the study will also compare CGM to conventional self-monitored blood glucose methods.

The study will also compare subjects' changes, if any, in nutrient intake such as energy, protein, fat and carbohydrate during the course of the study through interpretation/analysis of self-reported food intake.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (if of child-bearing age must practice appropriate birth control such as tubal ligation, oral contraceptives, abstinence or vasectomized partner during the duration of the study)
* Previously diagnosed with type 2 diabetes
* Age 21 and older
* Treated with metformin, a sulfonylurea, a thiazolidinedione, a combination or metformin and a sulfonylurea, or a combination of metformin and a thiazolidinedione (approved FDA indications)
* HbA1c 7.1-11%, unless subject has been using exenatide prior to study; in that case, there is no restriction on HbA1c level.
* Willing to give informed consent
* Motivated and capable of following the protocol and instructions provided by the healthcare professional
* Available for the study on the scheduled visit days
* Access to telephone communications

Exclusion Criteria:

* Under 21 years of age
* Pregnancy
* Creatinine clearance <30 ml/min (using MDRD formula)
* Known gastrointestinal disease
* Without diabetes or known type 1 diabetes
* Unable to follow the study protocol
* Unable to read and write in English
* Allergy to adhesives
* Any concomitant medical condition that would likely affect the evaluation of CGM device performance as determined by the investigator such as dermatological conditions or myxedema.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Mazze, PhD, Principal Investigator — International Diabetes Center - Park Nicollet Institute; Robert M. Cuddihy, MD, Principal Investigator — International Diabetes Center - Park Nicollet Institute; Ellie Strock, ANP, Principal Investigator — International Diabetes Center - Park Nicollet Institute
Locations (1):
- International Diabetes Center - Park Nicollet Health Services, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Mazze RS, Lucido D, Langer O, Hartmann K, Rodbard D. Ambulatory glucose profile: representation of verified self-monitored blood glucose data. Diabetes Care. 1987 Jan-Feb;10(1):111-7. doi: 10.2337/diacare.10.1.111. PMID 3552508
- [Background] Buse JB, Henry RR, Han J, Kim DD, Fineman MS, Baron AD; Exenatide-113 Clinical Study Group. Effects of exenatide (exendin-4) on glycemic control over 30 weeks in sulfonylurea-treated patients with type 2 diabetes. Diabetes Care. 2004 Nov;27(11):2628-35. doi: 10.2337/diacare.27.11.2628. PMID 15504997
- [Background] DeFronzo RA, Ratner RE, Han J, Kim DD, Fineman MS, Baron AD. Effects of exenatide (exendin-4) on glycemic control and weight over 30 weeks in metformin-treated patients with type 2 diabetes. Diabetes Care. 2005 May;28(5):1092-100. doi: 10.2337/diacare.28.5.1092. PMID 15855572
- [Background] Garg S, Zisser H, Schwartz S, Bailey T, Kaplan R, Ellis S, Jovanovic L. Improvement in glycemic excursions with a transcutaneous, real-time continuous glucose sensor: a randomized controlled trial. Diabetes Care. 2006 Jan;29(1):44-50. doi: 10.2337/diacare.29.01.06.dc05-1686. PMID 16373894